CLINICAL TRIAL: NCT02509962
Title: Effects of Increased Salt Intake on Metabolic, Cardiovascular and Immunoregulatory Functions in Healthy Men
Brief Title: Increased Salt Intake in Healthy Men
Acronym: BSALT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Anja Maehler, Principle Investigator, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Tissue Salt 3
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Energy metabolism; Glucose tolerance; Blood pressure; Immunoregulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Slow sodium tablets (Experimental): Increased dietary salt intake
  Interventions: Dietary Supplement: Slow sodium tablets

INTERVENTIONS:
Dietary Supplement: Slow sodium tablets — 6 g sodium chloride per day over 14 days

SUMMARY:
To study the effects of an increased salt intake on metabolic, cardiovascular and immunoregulatory functions in healthy men.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 18.5 - 29.9 kg/m2

Exclusion Criteria:

* clinically relevant heart, lung, liver, and kidney diseases

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Postprandial energy expenditure within 4h after a meal, measured by indirect calorimetry (respiratory chamber) | Change to baseline at day 14

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boschmann, Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Experimental & Clinical Research Center, Berlin, Germany

REFERENCES:
- [Result] Wilck N, Matus MG, Kearney SM, Olesen SW, Forslund K, Bartolomaeus H, Haase S, Mahler A, Balogh A, Marko L, Vvedenskaya O, Kleiner FH, Tsvetkov D, Klug L, Costea PI, Sunagawa S, Maier L, Rakova N, Schatz V, Neubert P, Fratzer C, Krannich A, Gollasch M, Grohme DA, Corte-Real BF, Gerlach RG, Basic M, Typas A, Wu C, Titze JM, Jantsch J, Boschmann M, Dechend R, Kleinewietfeld M, Kempa S, Bork P, Linker RA, Alm EJ, Muller DN. Salt-responsive gut commensal modulates TH17 axis and disease. Nature. 2017 Nov 30;551(7682):585-589. doi: 10.1038/nature24628. Epub 2017 Nov 15. PMID 29143823
- [Derived] Geisberger S, Bartolomaeus H, Neubert P, Willebrand R, Zasada C, Bartolomaeus T, McParland V, Swinnen D, Geuzens A, Maifeld A, Krampert L, Vogl M, Mahler A, Wilck N, Marko L, Tilic E, Forslund SK, Binger KJ, Stegbauer J, Dechend R, Kleinewietfeld M, Jantsch J, Kempa S, Muller DN. Salt Transiently Inhibits Mitochondrial Energetics in Mononuclear Phagocytes. Circulation. 2021 Jul 13;144(2):144-158. doi: 10.1161/CIRCULATIONAHA.120.052788. Epub 2021 Apr 28. PMID 33906377
- See also: Results publication — https://www.nature.com/articles/nature24628